CLINICAL TRIAL: NCT07345741
Title: Clinical Study on the Safety and Efficacy of CD20/CD19 Cell Injection in the Treatment of Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Donghua Zhang (Other)
Responsible Party: Sponsor-Investigator, Donghua Zhang, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHZ1962-E
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: R/R B-NHL; Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (R/R B-NHL)
Keywords: relapsed or refractory B-cell non-Hodgkin lymphoma (R/R B-NHL)
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:Experimental group (Experimental)
  Interventions: Drug: AcNK-Sup003 cell injection

INTERVENTIONS:
Drug: AcNK-Sup003 cell injection — AcNK-Sup003 cell injection in subjects with relapsed or refractory B-cell non-Hodgkin lymphoma (R/R B-NHL)

SUMMARY:
Evaluate the safety and tolerability of AcNK-Sup003 cell injection in subjects with relapsed or refractory B-cell non-Hodgkin lymphoma (R/R B-NHL). To preliminarily determine the Maximum Tolerated Dose (MTD) or recommended clinical dose of AcNK-Sup003 cell injection.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent: Signed written informed consent and ability to comply with protocol-specified visits and procedures.

Age and life expectancy: Age ≥ 18 years with an expected survival of more than 3 months.

Pathological diagnosis: Histopathologically confirmed CD20+ relapsed or refractory B-cell non-Hodgkin lymphoma (according to WHO 2016 lymphoma classification), including but not limited to:

Diffuse large B-cell lymphoma (DLBCL) High-grade B-cell lymphoma (HGBCL) Follicular lymphoma grade 3b (3b FL)

Relapsed or refractory disease: Defined by meeting one or more of the following:

Relapse, non-response, or progression after hematopoietic stem cell transplantation Stable disease for ≤ 6 months after at least two cycles of second-line therapy (DLBCL/HGBCL/3b FL subtypes must have received CD20-targeted agents and anthracyclines; other subtypes evaluated by investigator for treatment adequacy) Disease progression or relapse after at least second-line therapy (DLBCL/HGBCL/3b FL subtypes must have received CD20-targeted agents and anthracyclines; other subtypes evaluated by investigator for treatment adequacy) ECOG performance status: 0-2.

Contraception requirements:

Fertile males and females of childbearing potential must agree to use effective contraception from signing informed consent until 6 months after last study drug administration Negative serum pregnancy test required for females of childbearing potential at screening

Measurable disease: At least one measurable lesion according to Lugano 2014 criteria:

Lymph node lesions > 15mm in longest diameter on CT Extranodal lesions > 10mm in longest diameter FDG-PET positive (SUV ≥ 4 or 5) Radiated lesions only considered measurable if progression documented after completion of radiotherapy

Hematological parameters (no blood transfusion or hematopoietic growth factor within 7 days prior to testing):

Hemoglobin (Hb) ≥ 80 g/L Absolute neutrophil count (ANC) ≥ 1×10⁹/L Platelet count (PLT) ≥ 50×10⁹/L

Coagulation function:

International Normalized Ratio (INR) ≤ 1.5×ULN Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN (INR 2.0-3.0 acceptable for subjects on prophylactic anticoagulation)

Organ function requirements:

Renal: Serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula) Hepatic: Total bilirubin ≤ 1.5×ULN (≤ 3×ULN for liver infiltration or Gilbert's syndrome); ALT and AST ≤ 3×ULN (≤ 5×ULN for liver infiltration) Pulmonary: Oxygen saturation ≥ 92% on room air Subjects failing to meet any of the above criteria will not be eligible for enrollment.

Exclusion Criteria:

Primary CNS involvement: Primary central nervous system lymphoma or active CNS involvement/symptoms.

Autoimmune conditions: Active autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, autoimmune thrombocytopenia) or uncontrolled pleural effusions.

Cardiovascular history:

Severe cardiac rhythm/conduction abnormalities requiring intervention QTcF prolongation (> 450 ms males, > 470 ms females) Acute coronary syndrome, heart failure, aortic dissection, stroke, or other ≥ grade 3 cardiovascular events within 6 months NYHA class ≥ II heart failure or LVEF < 50% Uncontrolled hypertension (systolic ≥ 160 mmHg and/or diastolic ≥ 100 mmHg despite medication)

Prior cell therapies/transplants:

Autologous stem cell transplant or cell therapy within 3 months Allogeneic stem cell transplant or cell therapy within 6 months History of solid organ transplantation Prior anticancer therapy: Anticancer treatment or participation in other interventional clinical studies within 4 weeks or 5 half-lives (whichever is shorter) before lymphodepletion.

Recent procedures/vaccinations: Live attenuated vaccine or major surgery within 4 weeks before lymphodepletion, or planned during study.

Systemic steroids: Requirement for prolonged (≥ 3 days) systemic steroid therapy (≥ 10 mg/day prednisone equivalent) during study (inhaled or topical steroids excluded).

Other malignancies/conditions: History of other malignancies (except cured in-situ cervical cancer, non-invasive skin cancers, or locally treated prostate/breast carcinoma with ≥ 2 years remission); severe diabetes or other serious comorbidities.

Active infections: Active fungal, bacterial, viral, or mycobacterial infections requiring systemic treatment within 14 days before lymphodepletion.

Infectious diseases:

HBsAg positive or HBcAb positive with detectable HBV DNA HCV antibody positive with detectable HCV RNA HIV antibody positive Active syphilis Hypersensitivity: Life-threatening hypersensitivity or intolerance to study medications or severe allergic diathesis.

Pregnancy/lactation: Pregnant or breastfeeding females. Other factors: Any condition deemed by investigator to affect compliance or make subject unsuitable for study participation.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time frame:1, 3,6,12,18, 24 months after treatment
  Time frame:1, 3,6,12,18, 24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China